CLINICAL TRIAL: NCT07350941
Title: RAP-IC Study: Impact of Cardiac Rehabilitation Adapted for Patients With Heart Failure
Brief Title: Impact of Cardiac Rehabilitation Adapted for Patients With Heart Failure
Acronym: RAP-IC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Margarita Calvo López, Principal Investigator, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI 195/25
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac rehabilitation; Cardiopulmonary stress test; Functional capacity
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehabilitation group (treatment group) (Experimental): 3 months of a cardiac rehabilitation program, in which patients will attend in person twice weekly (Mondays and Wednesdays or Tuesdays and Thursdays), in groups of up to 8 patients, for 1-hour exercise sessions including aerobic, resistance, respiratory, and balance/proprioceptive components. Sessions will be monitored and supervised by cardiologists, rehabilitation physicians, and physiotherapists. In addition, patients will attend one weekly in-person educational session throughout the 3-month program.
  Interventions: Other: Cardiac rehabilitation program
- No intervention group (No Intervention): General exercise and educational recommendations

INTERVENTIONS:
Other: Cardiac rehabilitation program — Cardiac rehabilitation program, in which patients will attend in person twice weekly (Mondays and Wednesdays or Tuesdays and Thursdays), in groups of up to 8 patients, for 1-hour exercise sessions including aerobic, resistance, respiratory, and balance/proprioceptive components. Sessions will be monitored and supervised by cardiologists, rehabilitation physicians, and physiotherapists. In addition, patients will attend one weekly in-person educational session throughout the 3-month program.
  Arms: Cardiac rehabilitation group (treatment group)

SUMMARY:
The aim of the study is to evaluate whether a tailored cardiac rehabilitation program, initiated during hospitalization and continued after discharge, can improve functional capacity, mobility, and quality of life in patients over 65 years old with heart failure.

DETAILED DESCRIPTION:
If you meet the inclusion criteria and wish to participate, an initial assessment of your clinical and functional status will be conducted during your hospital stay. A computer system will then randomly assign you to one of the following groups:

Cardiac Rehabilitation Group (treatment group): You will participate in a mild exercise program during hospitalization (Phase I), including mobility and respiratory exercises adapted to your clinical condition. After discharge, you will enter a structured in-person cardiac rehabilitation program (Phase II) lasting 3 months, consisting of two 1-hour exercise sessions per week (aerobic, strength, inspiratory, and proprioceptive exercises) plus one weekly educational session.

Usual Care Group (control group): You will receive standard recommendations for physical activity and general care.

At the end of the study, a final consultation will be conducted to assess differences between the two groups in functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for acute heart failure in a stable phase (on a stable dose or tapering intravenous diuretics for at least 48 hours, without intravenous inotropes or vasodilators for >72 hours).
* Baseline functional class II-III
* Age ≥ 65 years
* Able to walk >4 meters
* Any range of left ventricular ejection fraction

Exclusion Criteria:

* Moderate to severe dementia
* Cardiac or other disease with a life expectancy <12 months
* Institutionalized patients or unable to travel to the rehabilitation center
* Functional class I or IV
* Uncontrolled arrhythmias
* Inability to perform a basic exercise protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: Change in Peak Oxygen Uptake | 3 months
  Change in peak oxygen uptake measured by treadmill cardiopulmonary exercise testing (peak VO₂, measured in ml/kg/min).

SECONDARY OUTCOMES:
Change in Functional Permormance assessed by the Short Physical Performance Battery (SPPB) score | 3 months
  Change in the Short Physical Performance Battery (SPPB) score, ranging from 0 (worst physical performance) to 12 (best physical performance).
Change in the Kansas City Cardiomyopathy Questionnaire-23 (KCCQ-23) score | 3 and 6 months
  Change in the Kansas City Cardiomyopathy Questionnaire-23 (KCCQ-23) overall summary score, ranging from 0 (worst health status) to 100 (best health status)
Change in distance walked (meters) in the 6-Minute Walk Test (6MWT). | 3 and 6 months
  Change in distance walked (meters) in the 6-Minute Walk Test (6MWT).
Change in caregiver burden assessed by the Zarit scale | 3 and 6 months
  Change in caregiver burden assessed by the 22-item Zarit Burden Interview (ZBI-22) score (range 0-88, with higher scores indicating greater caregiver burden)
Change in body composition parameters assessed by bioelectrical impedance analysis (BIA) | 3 and 6 months
  Change in body composition parameters expressed as percentages (%), assessed by bioelectrical impedance analysis (BIA)
Number of participants experiencing all-cause mortality, heart failure decompensation, or heart failure-related hospitalization during follow-up | 3 and 6 months
  All-cause mortality will be confirmed by medical records or death certificate. Heart failure decompensation will be defined as worsening of heart failure symptoms requiring urgent medical visit, treatment adjustment, or hospital admission. Heart failure-related hospitalizations will be collected from hospital records. Data will be aggregated as the number and percentage of participants experiencing each event during the study period
Change in Frailty status assessed by FRAIL scale | 3 and 6 months
  Change in FRAIL scale (range 0-5, higher scores indicate greater frailty)
Change in emotional status assessed by the Hospital Anxiety and Depression Scale (HADS) | 3 and 6 months
  Change in emotional status, measured using the Hospital Anxiety and Depression Scale (HADS), with subscales for anxiety and depression ranging from 0 to 21, where higher scores indicate greater symptom severity
Change in Nutritional Status assessed using the Mini Nutritional Assessment (MNA) score | 3 and 6 months
  Change in nutritional status, assessed using the Mini Nutritional Assessment (MNA) score (range 0-30, with higher scores indicating better nutritional status)
Change in Maximal Inspiratory Pressure (MIP) | 3 and 6 months
  Change in maximal inspiratory pressure (MIP) measured in cmH₂O, with higher values indicating greater respiratory muscle strength
Patient satisfaction | 6 months
  Patient satisfaction with the cardiac rehabilitation program, rated from 0 to 10, being 10 the highest mark
Patient adherence | 3 months
  Patient adherence to cardiac rehabilitation sessions, rated from 0 to 100%, being 100% the highest mark
Change in basic functional independence assessed by the Barthel Index | 3 and 6 months
  Change in basic functional independence assessed by the Barthel Index (range 0-100, with higher scores indicating greater independence)
Change in maximal expiratory pressure (MEP) | 3 ad 6 months
  Change in maximal expiratory pressure (MEP) measured in cmH₂O, with higher values indicating greater respiratory muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Calvo-LOpez, MD, Principal Investigator — Hospital Universitario Puerta de Hierro
Locations (1):
- Hospital Universitario Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial